CLINICAL TRIAL: NCT07336381
Title: An Exploratory Clinical Study Using the Replexa+ Device in Veterans With Lower Extremity Peripheral Artery Disease Experiencing Peripheral Neuropathy
Brief Title: Replexa+ Shortwave Diathermy Device for Patients Diagnosed With Peripheral Artery Disease and Peripheral Neuropathy
Acronym: Replexa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: ProMedTek, Inc. (Unknown)
Responsible Party: Principal Investigator, Michael Murphy, MD, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 29224
Record Dates: First submitted 2026-01-11; First posted 2026-01-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Arterial Disease; Peripheral Neuropathy
Keywords: peripheral artery disease; peripheral neuropathy; lower extremity artery disease; lower extremity neuropathy; PAD
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Experimental): In-home shortwave diathermy treatment.
  Interventions: Device: Replexa shortwave diathermy

INTERVENTIONS:
Device: Replexa shortwave diathermy — Treatment with home use of the Replexa+ shortwave diathermy device twice daily for 3 months.

SUMMARY:
This research project is designed to see if treatment with the Replexa+ shortwave diathermy device daily for 3 months will improve blood flow in the lower legs and feet of patients diagnosed with peripheral artery disease and peripheral neuropathy.

DETAILED DESCRIPTION:
This is a single-site, non-randomized, open label, exploratory clinical trial to evaluate the effects of the Replexa+ shortwave diathermy treatment in patients diagnosed with peripheral artery disease (PAD) and peripheral neuropathy. This pilot study will examine changes in lower extremity perfusion in a total of ten (10) Veteran patients at the Roudebush VA Medical Center in Indianapolis, Indiana, USA.

The proposed research will study the effects of the Replexa+ device, a Class II, non-invasive device that is cleared to market by the FDA (510k# K162240) and available to prescribing physicians at Veterans Affairs (VA) medical facilities. The Replexa+ device generates a form of electromagnetic energy (shortwave diathermy) to provide therapeutic heat to affected areas, deeper than infrared lights and heating pads. This type of therapeutic heat treatment has been widely used in clinical settings. The Replexa+ system consists of a generating unit (device) connected by a cable to a treatment applicator that is placed against the treated areas over normal clothing. The device operates at 27.12 megahertz (MHz), providing deep heating therapeutic effects to the body tissues.

Patients enrolled in this study will follow the manufacturer's instructions for use of the Replexa+ device and treatment. Treatment will comprise of two 30-minute sessions per day, approximately 8-12 hours apart, for 3 months, at prescribing physician-specified locations of the body.

At the post-treatment visit, the study doctor will assess the success or failure of treatment by comparing baseline measurement testing to post-treatment testing. Treatment failure will be defined as any measurable decrease in limb perfusion as evidenced by lower extremity arterial doppler testing.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of peripheral artery disease (PAD).
2. Participants must exhibit PAD severity, defined by the following manifestation and corresponding Rutherford classifications:

   Claudication of the index limb (Rutherford Category 2 or 3- documented as pain with walking) in conjunction with one or more of the following:
   * ankle brachial index (ABI) greater than or equal to 0.6 mmHg, as measured no more than 6 months prior to screening
   * resting toe brachial index (TBI) greater than or equal to 0.4, as measured no more than 6 months prior to screening

   Note: In cases where ankle and toe systolic pressures are unavailable due to calcification and/or toe amputation, collection of angiographic data is acceptable to determine locations of blockages or reduced perfusion.
3. Diagnosis of peripheral neuropathy, as evidenced by review of medical records.
4. Competent to give consent.
5. Age 18 years or older.

Exclusion Criteria:

1. Impaired skin integrity in the location(s) to be treated.
2. Current wounds or ulcerations.
3. Diagnosis of active bleeding tendencies, hemorrhage, or thrombosis.
4. 2+ pitting edema in either lower extremity.
5. Active infection defined as elevated white blood cell count >11,500/µL or fever >101.5 degrees Fahrenheit or currently taking antibiotic medication(s) for an active infection.
6. Existence of metal hardware in the area(s) to be treated: Any patient with implanted electronic or metal device such as a pacemaker, bladder stimulator, spinal cord stimulator or electrodes for a myoelectric prosthesis, IUD, surgical staples or implanted metallic leads.
7. Pregnant individuals.
8. Presence of renal disease (creatinine > 2.5 mg/dl and estimated glomerular filtration rate (eGFR) <30 mL/min) or patients on chronic hemodialysis.
9. History of skeletal tuberculosis.
10. Patients, in the investigator's opinion, whose index limb condition is rapidly deteriorating and may require major amputation within 30 days of screening.
11. Conditions that impair cognitive function.
12. Severe concomitant disease(s), or any additional condition(s) which the investigator feels constitute(s) criteria for exclusion of a particular subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare baseline and post-treatment lower extremity arterial dopplers to determine change in lower extremity arterial perfusion. | 3 months
  Patients will be treated twice daily for three months with the Replexa+ device. Lower extremity arterial dopplers (LEADs) will be assessed at baseline and post-treatment to determine improvement in lower extremity perfusion.

SECONDARY OUTCOMES:
Identify the presence and role of inflammatory biomarkers in PAD. | 3 months
  Patients will undergo peripheral blood collection at baseline and post-treatment time points to compare levels of high sensitivity C-reactive protein (hsCRP).

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Murphy, MD, Principal Investigator — VA Medical Center, Indiana University
Locations (1):
- Richard L. Roudebush Veterans Affairs Medical Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ProMedTek, Inc. website — http://promedtek.com
- See also: FDA 510(k) Premarket Notification — https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpmn/pmn.cfm?ID=K162240